CLINICAL TRIAL: NCT06180655
Title: An Integrative Online Diabetes Self-Management Education and Support Intervention Featuring Tai Chi Easy
Brief Title: Diabetes Self-Management Plus Tai Chi Easy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00003577
Record Dates: First submitted 2023-11-28; First posted 2023-12-22 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Self-Management; Tai Chi
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Palliative Care; Trichloroethylene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diabetes Self-Management Education and Support (DSMES) plus Tai Chi Easy (TCE)™ (Experimental): Participants will be asked to attend 45 minutes of DSMES and 45 min of TCE twice a week for 6 weeks. All classes will be recorded and available online and can viewed at a time when it is most convenient to accommodate working adults.
  Interventions: Behavioral: Diabetes Self-Management Education and Support (DSMES) plus Tai Chi Easy (TCE)™

INTERVENTIONS:
Behavioral: Diabetes Self-Management Education and Support (DSMES) plus Tai Chi Easy (TCE)™ — Participants will be asked to attend 45 minutes of DSMES and 45 min of TCE twice a week for 6 weeks. All classes will be recorded and available online and can viewed at a time when it is most convenient to accommodate working adults.

SUMMARY:
The purpose of this project is to increase access to diabetes care and education for adults aged 40-64 years old who are diagnosed with Type 2 Diabetes Mellitus and are unable to attend education and support classes due to their work situation. This project will use an established, well-known program for Diabetes Self-Management Education and Support (DSMES) and combine it with Tai Chi Easy (TCE)™ to enhance physical health, psychological health, and health behaviors. Participants will be asked to attend 45 minutes of DSMES and 45 min of TCE twice a week for 6 weeks. All classes will be recorded and available online and can viewed at a time when it is most convenient to accommodate working adults. Participants will be asked to complete survey questionnaires online, at the beginning and end of the program; and have a smart phone to connect with a smart ring during the 6-week DSMES+TCE program. After the program is done, participants will be asked to return the smart ring. Upon receipt of the smart ring, they will receive a give a gift card to thank them for their participation in the program.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with T2DM
* any sex/gender
* any race/ethnicity
* any socioeconomic group
* has a smartphone
* receives care in a Federally Qualified Healthcare Center in Southern Arizona

Exclusion Criteria:

* Individuals with T1DM
* Individuals with gestational DM
* Individuals with pre-diabetes
* children
* pregnant women
* Individuals unable to provide informed consent
* Individuals with other serious co-occurring health condition (e.g., active cancer treatment)

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Study Feasibility: Recruitment | screening pre-intervention
  the proportion of respondents who remained interested in the study after information and screening. Goal: recruit 10 participants per month for 3 months.
Study Feasibility: Retention | pre and post intervention at 6-weeks
  number of participants that completed all aspects of the study (data collection pre-post intervention and study intervention) Goal: 80% study retention
Study Feasibility: Intervention acceptability | post-intervention at 6-weeks
  The Acceptability of Intervention Measure (AIM) is brief and contains 4-items using a 5-point Likert scale (possible scores 4-20), with higher scores indicating greater acceptability of the intervention. Adequate reliability and validity have been reported. Benchmark: at least 75% intervention acceptability, across sites.
Study Feasibility: Intervention feasibility | post-intervention at 6-weeks
  The Feasibility of Intervention Measure (FIM) is brief and contains 4-items using a 5-point Likert scale (possible scores 4-20), with higher scores indicating greater feasibility of the intervention. Adequate reliability and validity have been reported. Benchmark: at least 75% intervention feasibility, across sites.
Study Feasibility: Intervention appropriateness | post-intervention at 6-weeks
  The Intervention Appropriateness Measure (IAM) is brief and contains 4-items using a 5-point Likert scale (possible scores 4-20), with higher scores indicating greater appropriateness of the intervention. Adequate reliability and validity have been reported. Benchmark: at least 75% intervention appropriateness, across sites.
Study Feasibility: Intervention safety | during the 6-week intervention
  number of adverse events during the intervention. Goal: no safety issues or adverse events

SECONDARY OUTCOMES:
self-reported physical health: Weight | pre-intervention (self-report)
  body weight in pounds
self-reported physical health: Height | pre-intervention (self-report)
  body height in inches
self-reported physical health: Waist Circumference | pre-intervention (self-report)
  waist circumference in inches
self-reported physical health: Blood Pressure | pre-intervention (self-report)
  blood pressure in millimeters of mercury (mm/Hg)
self-reported physical health: Blood Sugar | pre-intervention (self-report)
  blood sugar in milligrams per deciliter (mg/dL)
self-reported physical health: Hemoglobin A1C | pre-intervention (self-report)
  percentage of hemoglobin in blood that is coated with glucose
perceived psychological health: Diabetes Distress Scale | pre and post-intervention at 6-weeks
  The Diabetes Distress Scale (DSS-17) is a widely used, self-administered scale. The DDS-17 contains 17 items and asks a person about living with diabetes, using a six-point Likert format (1=not a problem, 6=a very serious problem). The DDS-17 contains questions related to emotional burden, physician distress, regimen distress and interpersonal distress. Possible scores range from 17 to 102, with higher scores indicating greater diabetes distress.
perceived psychological health: Patient Health Questionnaire-9 | pre and post-intervention at 6-weeks
  The Patient Health Questionnaire-9 (PHQ-9) is a widely used, self-administered scale to screen for depressive symptoms. The PHQ-9 contains 9 items that ask a person about problems that have been bothering them during the past 2 weeks, using a four-point Likert format (0=not at all, 3=nearly every day). Possible scores range from 0 to 27, with higher scores indicating greater severity of depressive symptoms.
perceived psychological health: Posttraumatic Stress Scale-Civilian Version | pre and post-intervention at 6-weeks
  The Posttraumatic Stress Scale-Civilian Version (PCL-C) is a self-administered scale that asks a person about problems or stressful life experiences during the past month. The PCL-C contains 17 items using a five-point Likert format (1=not at all, 5=extremely). Possible scores range from 17 to 85, with higher scores indicating greater symptoms associated with posttraumatic stress.
perceived psychological health: Diabetes Quality of Life Questionnaire | pre and post-intervention at 6-weeks
  The Diabetes Quality of Life Questionnaire (DQOL) is a self-administered scale that asks a person about their diabetes-related satisfaction, impact and worry. The DQOL contains 64 items using a using a five-point Likert format (satisfaction 1=very satisfied, 5=very dissatisfied; impact 1= no impact, 5=always impacted; worry 1=never worried, 5=always worried). Possible scores range from 64 to 320, with higher scores indicating worse quality of life.
perceived psychological health: Perceived Stress Scale | pre and post-intervention at 6-weeks
  The Perceived Stress Scale (PSS-10) is a widely used, self-administered scale. The PSS-10 contains 10 items and asks a person about situations they may have experienced in the past month as being unpredictable, uncontrollable, and overloaded using a five-point Likert format (0=never, 4=very often). Possible scores range from 0 to 40, with higher scores indicating greater perceived stress.
health behaviors: Dietary Screener Questionnaire | pre and post-intervention at 6-weeks
  The Dietary Screener Questionnaire (DSQ) is a 26-item self-administered scale that asks about the frequency of consumption of selected foods and drinks in the past month. The DSQ captures intakes of fruits and vegetables, dairy/calcium, added sugars, whole grains/fiber, red meat, and processed meat. The DSQ uses a scoring algorithm to convert responses to estimates of dietary intake for fruits and vegetables (cup equivalents), dairy (cup equivalents), added sugars (tsp), whole grains (ounce equivalents), fiber (g), and calcium (mg). Responses to the red meat and processed meat questions are as qualitative indicators of intake frequency, but no scoring algorithms were developed for those particular dietary factors.
health behaviors: Rapid Assessment of Physical Activity | pre and post-intervention at 6-weeks
  The Rapid Assessment of Physical Activity (RAPA) questionnaire is a widely used, self-administered scale to assess a person's engagement in physical activity during the week. The RAPA contains 9 yes/no questions. The first 7 questions assess weekly physical activity during free time (RAPA 1). Affirmative responses are reviewed to determine the person's level of physical activity during the week (1=sedentary, 7=active). Possible scores range from 1 to 7, with higher scores indicating greater the level and intensity of the physical activity. The last two questions include strength training and flexibility items (RAPA 2), which are scored separately (0=none, 1=strength training, 2=flexibility, 3=both). Possible scores range from 0 to 3, which indicate if the person is engaging in strength and flexibility exercise during the week.
Objective measures using an Oura Ring: Sleep | during the 6-week intervention
  Daily total sleep in hours and minutes
Objective measures using an Oura Ring: Physical Activity | during the 6-week intervention
  Daily total physical activity in number of steps
Objective measures using an Oura Ring: Heart Rate Variability | during the 6-week intervention
  Daily average heart rate variability during the night in milliseconds

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona College of Nursing, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
this is a feasibility study